CLINICAL TRIAL: NCT00345566
Title: Effect of the Protein Composition on the Gastric Emptying Rate in Children With Cerebral Paresis
Brief Title: Effect of Protein Composition on Gastric Emptying
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Numico Europe (Unknown)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UUSKBK28200706
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2006-06-28 (Estimated); Status verified 2006-06

CONDITIONS: Cerebral Palsy; Gastric Dysmotility; Enteral Feeding
Keywords: cerebral palsy; protein composition; gastric emptying rate; tube feeding
MeSH Terms: conditions — Cerebral Palsy

INTERVENTIONS:
Procedure: Nutrition composition

SUMMARY:
The protein composition of nutrition may affect the rate of gastric emptying and gastric fysiology. This is espesially important in children with neurologic impariment, who commonly rely on tube feedings, have feeding problems, nausea, vomiting, gastroesophageal reflux and delayed gastric emptying. We aim to find out whether 4 different protein sources affect the rate of gastric emptying and electrofysiology in this group of children.

DETAILED DESCRIPTION:
Several factors in nutrition are known to affect gastric emptying rate, such as energy content, temperature, viscosity etc. In infants the protein composition affects gastric emptying. Children with cerebral pasly commonly have foregut dysmotility - with nausea, vomiting, feeding intolerance and gastroesophageal reflux. Tube feedings, usually based on cows milk are commonly used.

Our hypothesis is that the source and thus protein composition of feeding affects gastric emptying rate and electrofysiology.

Using four different tube feedings, standardized for content of fat, glucose and calories, we will measure gastric emptying rate using C13 octanoic acid as well as electrogastrography will be recorded. The protein modules are derived from casein, whey/casein mixture, hydrolyzed whey and aminoacids. Children with cerebral paresis and gastrostomy will be included. Each serves as his / her own control.

The primary endpoint is gastric emptying rate, the secondary endpoint electrogastrography.

ELIGIBILITY:
Inclusion Criteria: Cerebral paresis, user of tube feedings through gastrostomy -

Exclusion Criteria: Use of valproic acid (interferes with breath test). Age >16 y.

-

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25
Dates: Start 2006-08; Study Completion 2007-12

PRIMARY OUTCOMES:
Gastric emptying, measured by octanoic acid breath test.

SECONDARY OUTCOMES:
Electrogastrography

CONTACTS AND LOCATIONS:
Overall Officials: Ketil Stordal, PHD, Study Chair
Locations (1):
- Ullevaal university hospital, Oslo, Norway

REFERENCES:
- [Derived] Brun AC, Stordal K, Johannesdottir GB, Fossum V, Bentsen BS, Medhus AW. Nissen fundoplication in children with cerebral palsy: influence on rate of gastric emptying and postprandial symptoms in relation to protein source in caloric liquid meals. Clin Nutr. 2013 Aug;32(4):619-23. doi: 10.1016/j.clnu.2012.11.010. Epub 2012 Nov 17. PMID 23196118